CLINICAL TRIAL: NCT04516668
Title: Survey About Anxious and Depressive Symptoms During COVID-19 in Women Who Have Medical History of Post-partum Depression: Interest of Tele-consultation
Brief Title: Effect of Tele-consultation in Addition With Psychiatric Follow-up During COVID-19 in Women Who Have Medical History of Post-partum Depression
Acronym: COVIDDEPERINAT
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP200878
Record Dates: First submitted 2020-08-17; First posted 2020-08-18 (Actual); Last update posted 2020-10-06 (Actual); Status verified 2020-07

CONDITIONS: Post Partum Depression
Keywords: Post Partum Depression; Tele-consultation; COVID-19
MeSH Terms: conditions — Depression, Postpartum; COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Women who were able to benefit from psychiatric follow-up during the quarantine by tele-consultation have a lower risk of anxious and depressive symptoms than those who did not receive follow-up.

DETAILED DESCRIPTION:
The pandemic of COVID-19 (coronavirus desease 19) led to a strict quarantine from 15 March 2020 to 11 May 2020. Maternal depression is a current pathology , especially in the post-partum (more than 15%). The quarantine could lead to anxious and/or depressive symptoms and difficulties in parents-children bonding.

Women who have experenced post-partum period have more chance to developp subsequent depression.

Among women who have experienced post-partum depression, those who were able to benefit from psychiatric follow-up during the quarantine by tele-consultation have a lower risk of anxious and depressive symptoms than those who did not receive follow-up.

ELIGIBILITY:
Inclusion Criteria:

Women above 18 years old

Who have experienced a post-partum depression between 2013 and late of 2019

Who have benefit a psychiatry post-partum follow-up (hospitalizations in psychiatry post-partum unity and/or medical consultation) by Bicêtre psychiatry service

Who have a child less than 7 years old (preschool age)

Speaking and reading in french

And their partner (above 18 years old)

In the main analyze, only women with a indication of following psychiatric follow-up by tele-consultation (with a psychiatric follow-up at the begenning of the quarantine, who have not been follow-up by psychiatrist in hospitalization or in face to face consultation) will be analyzed

Exclusion Criteria:

People with chronic psychotic disorder (Diagnostic and Statistical Manual of Mental Disorders:DSM-5 criteria)

People with mental handicap

People who are not able to give their consent

People subject to protection measure

People refusing to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women who were treated by the psychiatry department at Bicêtre hospital for post-partum depression between 2013 and late 2019 and their partner
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2020-11 (Estimated); Primary Completion 2020-11 (Estimated); Study Completion 2020-11 (Estimated)

PRIMARY OUTCOMES:
Evaluation of Hospital anxiety and depression scale (HAD) | 15 minutes
  To compare depression and anxiety HAD score of women who have a medical history ofpost-partum depression according to a follow-up or not during the quarantine by tele-consultation
  Score less than or egal to 7 = no case Score between 8 and 10 = uncertain case Score higher than or equal to 11 = confirmed case

SECONDARY OUTCOMES:
Evaluation of Edinburgh Postpartum Depression Scale (EPDS) | 15 minutes
  To compare the result of EPDS in women who have a child of less 2 years old according to a follow-up or not by tele-consultation during the quarantine
Evaluation of HAD score in fathers | 15 minutes
  Anxiety and depression of fathers will be assessed with HAD scale
Evaluation of EPDS in fathers | 15 minutes
  EPDS will be assessed in fathers who have a child of less than 2 years old
Study of the relationship between maternals and paternals symptoms | 15 minutes
  The aim is to show that maternals anxious and depressive symptoms would be correlated to paternals positively symptoms
Study of difficuties in child during the quarantine | 15 minutes
  Look for a correlation between the difficulties in child during the quarantine describe by parents and anxiety and depression symptoms in parents The difficulties in child will be illustrated with the rate of children with difficulties describe by the parents
Risk and protection factors | 15 minutes
  Description of risk factors and protection factors setting up by the family during this quarantine period

CONTACTS AND LOCATIONS:
Overall Officials: Florence Gressier, Dr, Principal Investigator — Bicêtre Hospital